CLINICAL TRIAL: NCT01528358
Title: Tissue NIRS in the Assessment and Management of Critically Ill Patients
Brief Title: Tissue Near InfraRed Spectroscopy (NIRS) in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, John Murkin, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Other Study IDs: R11375
Record Dates: First submitted 2012-02-02; First posted 2012-02-08 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Sepsis; Inflammation; Shock
Keywords: sepsis; tissue oximetry; NIRS; VOT
MeSH Terms: conditions — Sepsis; Inflammation; Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood: inflammatory markers
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early Sepsis Critically Ill Patients: Patients who are admitted to ICU with a diagnosis of early sepsis.
- Non-septic Critically ill patients: Patients who are critically ill and admitted to ICU without diagnosis of sepsis.

SUMMARY:
Hypotheses:

1. In the acute phase of early illness, tissue oxygen saturation and vascular occlusion test (VOT) are important adjuncts in differentiating severe critical illness requiring ICU admission from patients benefiting from less aggressive therapies (non-ICU admission).
2. An early feature of severe sepsis is abnormal microcirculatory vasoreactivity.
3. Microvascular reactivity can be measured by means of vascular occlusion test (VOT) using non-invasive near infrared spectroscopy (NIRS) to measure tissue Oxygen saturation (StO2).
4. Microvascular reactivity is significantly deranged in patients with early severe sepsis and is quantifiably different from non-septic critically ill patients.
5. Other measures of microcirculatory perfusion ie. sublingual orthogonal polarization spectral (OPS) video microscopy, are abnormal and will directionally correlate with VOT and StO2 in severe sepsis
6. In severely septic patients response to therapy can be assessed by VOT and StO2 monitoring and will correlate with prognosis.
7. A management protocol incorporating VOT and StO2 monitoring in addition to conventional hemodynamic and biochemical parameters as a guide to therapy will result in improved outcomes in severely septic patients.

This project will investigate the use of a non-invasive near infrared light (NIR) device in conjunction with brief arm compression to measure the microcirculation in critically ill patients. It is know that in patients with overwhelming infections, their blood vessels do not respond normally and the NIR device can help measure how abnormal their blood vessels are. This type of testing is non-invasive and can be performed repeatedly without harm to the patient and may provide an earlier way to determine whether they have overwhelming sepsis and also may help to optimize the treatments they receive and better tailor their treatments to the degree of blood vessel abnormalities that are found. If our hypotheses are correct, this simple non-invasive test could provide a very rapid means of assessing patients that could be done more safely and quickly than some of the current methods. This would have an important effect to enhance patient safety and improve outcomes in such critically ill patients.

DETAILED DESCRIPTION:
Project Overview: This project is focused on the early diagnosis and management of septic shock using tissue near infrared spectroscopy (tNIRS) for continuous and non-invasive assessment of microcirculatory vasoreactivity as a diagnostic and prognostic indicator in critically ill patients. A novel aspect of this study is that point of entry of patients will be via the Critical Care Outreach Team (CCOT) which will ensure patients are assessed in the early phases of their disease prior to and co-incident with admission to Critical Care Unit (CCU). The investigators will employ tNIRS to assess peripheral tissue oxygen saturation (StO2) in all patients assessed by CCOT (n = 1031 patients in 2009) and in addition, the investigators will employ the NIRS vascular occlusion test (VOT) using a brief episode of forearm ischemia to quantify microvascular (dys)function.

All patients admitted to CCU via CCOT (n = 230 patients in 2009) will have StO2 monitored and VOT assessment sequentially throughout the course of their critical illness. Biomarkers to assess severity of illness, inflammatory processes and microcirculatory reactivity will be obtained, and in a subset of patients (n = 30), correlations between these parameters and other indices of microvascular perfusion using sublingual orthogonal polarization spectral (OPS) imaging videomicroscopy will be sought. As it is estimated that 20-30% of CCOT admissions are for sepsis (n = 40-60), the inclusion of other critically ill non-septic patients will enable discrimination of various parameters of VOT to be contrasted between groups to determine relative diagnostic and prognostic significance.

Statement of Objectives:

1. To assess the diagnostic utility of tNIRS StO2 and VOT in early assessment of critically ill patients.
2. To determine whether significant and pathognomonic differences exist in StO2 and indices of VOT between septic patients versus other non-septic critically ill patients and healthy age matched volunteers.
3. To determine whether correlations exist between biomarkers of inflammation and vasoreactivity and measures of StO2 and VOT in severely septic patients.
4. To determine whether incorporation of StO2 and VOT into a treatment protocol can positively impact clinical outcomes in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing assessment by critical care outreach team.

Exclusion Criteria:

* non-consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients early in clinical course of illness.
Sampling Method: Non-Probability Sample
Enrollment: 672 (Actual)
Dates: Start 2012-04-04 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
tNIRS Reperfusion slope of VOT | 12 months
  Sequential mesures of tNIRS VOT will be performed in septic and non-septic patients early in thier clinical course and reperfusion slope of VOT will be contrasted between these patient groups.

SECONDARY OUTCOMES:
tNIRS for Management of Critically Ill Patients with Sepsis | 12 months
  In second phase of study patients critically ill with sepsis will be randomized to either use or non-use of tNIRS and VOT as a component of their clinical management. Number of survivors, length of ICU stay, SOFA and Apache scores on discharge from ICU will be compared between patients with either use or non-use of VOT-derived reperfusion slope which will be employed as a guide to monitor adequacy of tissue microcirculation and response to therapy.

CONTACTS AND LOCATIONS:
Overall Officials: John Murkin, MD, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- University Hospital, London Health Sciences Center, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided